CLINICAL TRIAL: NCT03431220
Title: A Prospective, Non-Comparative, Open, Multi-Center Study to Assess the Use of a New Negative Pressure Wound Therapy (NPWT) System (RENASYS Touch and RENASYS AB) in Temporary Abdominal Closure (TAC) For the Management of the Open Abdomen
Brief Title: Non-Comparative Study of Open Abdomen That Require the Use of Negative Pressure Wound Therapy (NPWT) for Temporary Abdominal Closure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 305-001-001-01
Record Dates: First submitted 2016-11-17; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Abdomenal Wound Trauma
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RENASYS TOUCH NPWT System (Experimental): Negative Pressure Wound Therapy (NPWT)
  Interventions: Device: RENASYS® TOUCH Negative Pressure Wound Therapy (NPWT) Device

INTERVENTIONS:
Device: RENASYS® TOUCH Negative Pressure Wound Therapy (NPWT) Device — NPWT applied to Grade 1 or Grade 2 open abdomen wounds for temporary abdominal closure for up to 14 days, with a 21 day post study initiation follow-up assessment.

SUMMARY:
A study in which subjects with a Grade 1 or Grade 2 open abdomen that require the use of NPWT for temporary abdominal closure. Subjects will use the NPWT system for up to 14 days, with a 21 day post study initiation follow-up assessment for latent complications and mortality.

ELIGIBILITY:
INCLUSION CRITERIA

1. Eligible subjects must be properly consented before enrollment. If the subject is incapable of providing consent, emergency consent procedures will be followed, or the subject's legal representative must be asked to provide consent on the subject's behalf, per the IRB guidelines.
2. Subjects must be at least eighteen (18) yeaTS of age, or older.
3. Males and non-pregnant females.
4. Grade 1 or Grade 2 open abdomen patients who would benefit from temporary abdominal closure (TAC) with topical Negative Pressure Wound Therapy (NPWT).

EXCLUSION CRITERIA

1. Grade 3 and Grade 4 open abdomens.
2. Malignancy in the reference wound bed or margins of the wound.
3. Patients with non-enteric unexplored fistulas.
4. High risk for imminent death, as determined by the attending surgeon and Principal Investigator (PI).
5. Pre-existing large ventral hernia.
6. Significant loss of abdominal wall fascia as a result of trauma or infection.
7. Patients with a known hist01y of poor compliance with medical treatment.
8. Patients who have participated in this trial previously and who were withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To determine the number of days taken to achieve delayed primary fascial closure. | 14 days
  NPWT applied to Grade 1 or Grade 2 open abdomen wounds for temporary abdominal closure for up to 14 days, with a 21 day post study initiation follow-up assessment.

SECONDARY OUTCOMES:
To confirm the performance of the NPWT system in terms of maintenance of abdominal tissue domain | 14 days
To confirm the performance of the NPWT system in terms of: management of peritoneal fluid | 14 days
To confirm the performance of the NPWT system in terms of reduction in edema | 14 days
To confirm the performance of the NPWT system in terms of prevention of fixity | 14 days
To confirm the performance of the NPWT system in terms of prevention of infection | 14 days
To assess the ability of the NPWT system to prevent further deterioration of the open abdomen as classified by Bjorck et al., (2009) | 14 days
To determine the type (method) of final closure of the open abdomen | 14 days
To assess the number of days to achieve final closure of the open abdomen | 14 days
To monitor the length of stay (days) in ICU and length of stay in hospital | 14 days
To monitor the number and type of re-operations throughout the course of the study | 14 days
To assess the number of dressing changes | 14 days
To record clinicians' overall opinion on the usability of the new device throughout the study | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jaime E Dickerson, PhD, Study Chair — Smith & Nephew, Inc.
Locations (1):
- Chicago, Illinois, United States